CLINICAL TRIAL: NCT01680965
Title: Ofatumumab in Combination With Glucocorticoids for Primary Therapy of Chronic Graft Versus Host Disease
Brief Title: Ofatumumab as Primary Therapy of Chronic Graft Versus Host Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-17071
Record Dates: First submitted 2012-09-04; First posted 2012-09-07 (Estimated); Results first posted 2020-11-12 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-09

CONDITIONS: Chronic Graft Versus Host Disease
Keywords: Graft vs. Host Disease; GVHD; chronic graft versus host disease (cGVHD); Allogeneic Transplant; Ofatumumab
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Graft vs Host Disease | interventions — ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ofatumumab (Experimental): Phase I:
  Escalating dose of ofatumumab
  Phase II:
  Maximum tolerated dose (MTD) of Ofatumumab
  Interventions: Drug: Ofatumumab

INTERVENTIONS:
Drug: Ofatumumab — Phase I: test an escalating dose of ofatumumab at cohorts of 300 mg, 700 mg, and 1000 mg given on day 0 and 14 of study.
  Phase II: Ofatumumab MTD on day 0 and 14; patients will be followed for total of 24 months (months 1, 3, 6, 12 after therapy, then at 18 and 24 months following therapy)

SUMMARY:
To study the safety and side effects of Ofatumumab in the treatment of chronic graft-versus-host disease (GvHD). This study will also evaluate effectiveness of Ofatumumab when added to standard steroid treatment for chronic graft-versus-host disease

DETAILED DESCRIPTION:
This is a phase I-II trial to examine the safety and efficacy of prednisone and escalating dose of ofatumumab for the primary therapy of chronic GVHD.

ELIGIBILITY:
Inclusion Criteria:

* Hematopoietic cell transplantation (HCT) recipients newly requiring systemic glucocorticoid therapy (at ≥ 1mg/kg/day prednisone or equivalent) for chronic GVHD
* Participants can be enrolled and begin study therapy with ofatumumab within 14 days from initiation of 1 mg/kg/day prednisone for therapy of chronic GVHD.

Exclusion Criteria:

* Relapse of primary hematologic malignancy that served as indication for HCT.
* Previous systemic glucocorticoid therapy (at ≥ 1mg/kg/day prednisone or equivalent) for chronic GVHD
* Prior systemic glucocorticoid therapy for acute GVHD is permitted
* Prior or ongoing systemic immune suppressive agents (including, but not limited to common examples such as calcineurin inhibitors, sirolimus, mycophenolate mofetil) provided for either prevention or treatment of acute GVHD are permitted and part of routine standard of care
* Current active hepatic or biliary disease (with exception of liver disease secondary to chronic GVHD, or patients with Gilbert's syndrome, asymptomatic gallstones, or stable chronic liver disease per investigator assessment).
* Patients with abnormal liver function tests due to chronic GVHD are specifically not excluded from the study. This is a common manifestation of chronic GVHD, and thus a major target for the study therapy.
* Treatment with experimental non-FDA approved therapy within 5 terminal half lives or 4 weeks prior to enrollment, whichever is longer
* Other past or current solid tumor malignancy
* Have been free of malignancy for at least 5 years, or have a history of completely resected non-melanoma skin cancer, or successfully treated in situ carcinoma are eligible.
* Prior treatment with anti-cluster of differentiation antigen 20 (CD20) monoclonal antibody or alemtuzumab within 3 months prior to start of therapy.
* Uncontrolled infectious complications not responsive to appropriate antimicrobial therapy.
* History of significant cerebrovascular disease (i.e. stroke or TIA) in the past 6 months or ongoing event with active symptoms or sequelae
* HIV positivity
* Uncontrolled, current significant cardiac disease including unstable angina, acute myocardial infarction within six months prior to randomization, congestive heart failure (NYHA III-IV), and arrhythmia unless controlled by therapy, with the exception of extra systoles or minor conduction abnormalities.
* A history of cardiac disease, such as coronary disease, arrhythmia or congestive heart failure that are on appropriate medical therapy and without evidence of current decompensation are eligible.
* Significant concurrent, uncontrolled medical condition including, but not limited to, renal, hepatic, gastrointestinal, endocrine, pulmonary, neurological, cerebral or psychiatric disease which in the opinion of the investigator may represent a risk for the patient.
* Those patients with medical conditions that are controlled with medical therapy are eligible.
* Clinically active Hepatitis B defined as positive HBsAg; or positive HBcAb with detectable hepatitis B virus (HBV) DNA viral load. Patients who are HBcAb with undetectable HBV DNA viremia are eligible.
* Positive serology for hepatitis C (HC) defined as a positive test and confirmed by HC recombinant immunoblot assay (RIBA) or hepatitis C virus (HCV) RNA viral load
* Screening laboratory value exclusion criteria: platelets < 50 x 10^9/L (patients with platelet counts > 50 x 10^9/L supported by platelet transfusion are eligible); neutrophils < 1.0 x 10^9/L (patients with an absolute neutrophil count > 1.0 x 10^9/L supported by growth factors are eligible); creatinine > 2.0 times upper normal limit; total bilirubin >1.5 times upper normal limit (unless due to chronic GVHD); alanine transaminase (ALT) > 2.0 times upper normal limit (unless due to chronic GVHD); alkaline phosphatase > 2.5 times upper normal limit (unless due to chronic GVHD).
* Women who are pregnant or lactating. Women of childbearing potential must have a negative pregnancy test at screening.
* Women of child bearing potential must undergo pregnancy testing within 7 days of the first dose of study therapy. Women must also undergo pregnancy test at 6 months after the last dose.
* Women of childbearing potential, including women whose last menstrual period was less than one year prior to screening, unable or unwilling to use adequate contraception from study start to one year after the last dose of protocol therapy. Adequate contraception is defined as hormonal birth control, intrauterine device, double barrier method or total abstinence.
* Males unable or unwilling to use adequate contraception methods from study start to one year after the last dose of protocol therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-11-14 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2020-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Pidala, MD, MS, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (4):
- United States (4):
  - Mayo Clinic Cancer Center, Phoenix, Arizona
  - H.Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - University of Minnesota, Minneapolis, Minnesota
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

REFERENCES:
- [Derived] Lazaryan A, Lee S, Arora M, Kim J, Betts BC, Khimani F, Nishihori T, Bejanyan N, Liu H, Kharfan-Dabaja MA, Locke FL, Gonzalez R, Jain MD, Davila ML, Perez LE, Mishra A, Perez Perez A, Balke K, Ayala E, Ochoa L, Castaneda Puglianini O, Faramand R, Alsina M, Elmariah H, Nieder ML, Fernandez H, Anasetti C, Pidala JA. A phase 2 multicenter trial of ofatumumab and prednisone as initial therapy for chronic graft-versus-host disease. Blood Adv. 2022 Jan 11;6(1):259-269. doi: 10.1182/bloodadvances.2021005552. PMID 34649279
- See also: H.Lee Moffitt Cancer Center & Research Institute — http://www.moffitt.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1 Cohort 1:Ofatumumab: Phase I Cohort 1: dose of ofatumumab at 300 mg given on day 0 and 14 of study.
- Phase 1 Cohort 2: Ofatumumab: Phase I Cohort 2: dose of ofatumumab at 700 mg given on day 0 and 14 of study.
- Phase1 Cohort 3: Phase I Cohort 3: dose of ofatumumab at 1000 mg given on day 0 and 14 of study.
- Phase 2: Maximum Tolerated Dose of Ofatumumab: Phase II: Maximum tolerated dose (MTD) of Ofatumumab
  Ofatumumab at 1000 mg on day 0 and 14
Period: Overall Study
Arm/Group | Phase 1 Cohort 1:Ofatumumab | Phase 1 Cohort 2: Ofatumumab | Phase1 Cohort 3 | Phase 2: Maximum Tolerated Dose of Ofatumumab
Started | 3 | 3 | 6 | 32
Completed | 3 | 3 | 6 | 26
Not Completed | 0 | 0 | 0 | 6
Not completed — Death | 0 | 0 | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Phase 1 Cohort 1: Ofatumumab: Phase I Cohort 1: dose of ofatumumab at 300 mg given on day 0 and 14 of study.
- Phase 1 Cohort 3: Ofatumumab: Phase I Cohort 3: dose of ofatumumab at 1000 mg given on day 0 and 14 of study.
- Total: Total of all reporting groups
Arm/Group | Phase 1 Cohort 1: Ofatumumab | Phase 1 Cohort 2: Ofatumumab | Phase 1 Cohort 3: Ofatumumab | Phase 2: Maximum Tolerated Dose of Ofatumumab | Total
Number analyzed (Participants) | 3 | 3 | 6 | 32 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 4 | 22 | 32
  >=65 years | 0 | 0 | 2 | 10 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3 | 10 | 16
  Male | 2 | 1 | 3 | 22 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 3 | 5
  Not Hispanic or Latino | 3 | 2 | 5 | 29 | 39
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 3 | 3 | 6 | 30 | 42
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6 | 32 | 44

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Ofatumumab
Description: Maximum Tolerated Dose was determined by increasing doses, beginning at 300 mg on day 0 and day 14, then increasing to 700 mg on day 0 and day 14 and finally 1000 mg on day 0 and day 14.
Time Frame: within 21 days of initiation
Population: All participants in phase 1 portion of study
Measure: Number; unit: mg
Groups:
- Phase 1: All Participants: All participants in phase 1 portion of study who received at least 1 dose of Ofatumumab either at 300 mg, 700 mg or 1000 mg.
Arm/Group | Phase 1: All Participants
Number analyzed (Participants) | 12
mg | 1000

2. Primary Outcome: Participants Response Rates
Description: Overall response rate (ORR) at 6 months following initiation of therapy. ORR is the composite outcome of complete response and partial response
Time Frame: 6 months following initiation of Ofatumumab
Population: Participants enrolled in Phase 2 portion of study
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Ofatumumab: Phase I:
  Escalating dose of ofatumumab
  Phase II:
  Maximum tolerated dose (MTD) of Ofatumumab
  Ofatumumab: Phase I: test an escalating dose of ofatumumab at cohorts of 300 mg, 700 mg, and 1000 mg given on day 0 and 14 of study.
  Phase II: Ofatumumab MTD on day 0 and 14; patients will be followed for total of 24 months (months 1, 3, 6, 12 after therapy, then at 18 and 24 months following therapy)
Arm/Group | Ofatumumab
Number analyzed (Participants) | 32
percentage of participants | 62.5 [44 to 79]

3. Secondary Outcome: Overall Survival (OS) at 24 Months
Description: Overall Survival is defined as the time period from start of treatment to death.
Time Frame: Up to 24 months
Population: Participants enrolled in Phase 2 portion of study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ofatumumab
Number analyzed (Participants) | 32
percentage of participants | 74.4 [56.6 to 85.8]

ADVERSE EVENTS:
Time Frame: 6 years, 6 months
Groups:
- Phase 1 Cohort 1: Phase I Cohort 1: dose of ofatumumab at 300 mg given on day 0 and 14 of study.
- Phase 1 Cohort 2: Phase I Cohort 2: dose of ofatumumab at 700 mg given on day 0 and 14 of study.
- Phase 1 Cohort 3: Phase I Cohort 3: dose of ofatumumab at 1000 mg given on day 0 and 14 of study.
- Phase 2: MTD: Phase II: Maximum tolerated dose (MTD) of Ofatumumab Ofatumumab at 1000 mg on day 0 and 14
Arm/Group | Phase 1 Cohort 1 | Phase 1 Cohort 2 | Phase 1 Cohort 3 | Phase 2: MTD
All-Cause Mortality (participants affected / at risk) | 2/3 | 1/3 | 3/6 | 9/32
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 4/6 | 25/32
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6 | 24/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Cohort 1 (N=3) | Phase 1 Cohort 2 (N=3) | Phase 1 Cohort 3 (N=6) | Phase 2: MTD (N=32)
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Lung Infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 3 (6)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Skin Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotrasnferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gallbladder obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders -Other (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periorbital edema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Surgical and medical procedures - Other (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Cohort 1 (N=3) | Phase 1 Cohort 2 (N=3) | Phase 1 Cohort 3 (N=6) | Phase 2: MTD (N=32)
Neutrophil Count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Diaphoresis
Infusion related reactions (General disorders) | 0 (0) | 1 (1) | 2 (2) | 8 (10)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower GI hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomach cramps (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper GI hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General disorders and administration site conditions -Other (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Fluid overload
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 4 (5)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (6)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal and urinary disorders - Other (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Dysuria
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Atrial fibrilation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other (Infections and infestations) | 1 (3) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (2) | 0 (0) | 2 (3) | 4 (4)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorders -Other (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — shakiness
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — wrist pain
Facial nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — coag negative staph in left hip incision
Vascular disorders - Other (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Surgical and medical procedures -Other (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 | 1 (1) — paraesophageal hernia repair
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders -Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Bronchial inflammation
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Staphylococcus
Bladder infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-10): https://cdn.clinicaltrials.gov/large-docs/65/NCT01680965/Prot_SAP_000.pdf